CLINICAL TRIAL: NCT00116051
Title: A Comparison of Two Surface Materials (Tantalum Versus Titanium Fiber Mesh) of Acetabular Components in Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Professor Kjeld Soballe, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Aarhus C
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200330159
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
Keywords: RSA; DEXA; Osteoarthritis; Hip arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Acetabular implant, Monoblock cup

SUMMARY:
The purpose of this study is to compare two surface materials (tantalum versus titanium fiber mesh) of acetabular components in hip arthroplasty.

DETAILED DESCRIPTION:
In younger patients, acetabulum components are most often implanted without the use of cement. A direct ingrowth of bone to the implant is crucial to the attainment of good results in those cases where cement is not employed. A new implant material (tantalum) has shown better properties than the implant material which is in use today (titanium). The advantages of tantalum implants are greater porosity, reduced stiffness and a higher friction coefficient than with titanium implants.

Hypothetically, the higher porosity of tantalum should enhance bone ingrowth due to better osteoconductivity in terms of:

1. less migration of the acetabulum component, as evaluated by RSA;
2. increased BMD in the bone surrounding acetabulum components;
3. fewer postoperative complaints on the Harris Hip Score and visual analog scale scores.

The migration of acetabulum components will be evaluated by RSA. The follow-up RSA will be scheduled for week 1, as well as 3 months, 12 months and 2 years after surgery. Bone mineral density around the implanted femoral component will be examined by DEXA scan at week 1, as well as 1 year and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary arthritis in the hip.
* Patients with sufficient bone density to allow uncemented implantation of a femoral component.
* Informed patient consent in writing.

Exclusion Criteria:

* Patients with neuromuscular or vascular disease in the affected leg.
* Patients found upon operation to be unsuited for uncemented acetabulum component.
* Patients who regularly take non-steroid anti-inflammatory drugs (NSAID) and cannot interrupt intake for the postoperative phase of the study.
* Patients with fracture sequelae.
* Female patients of childbearing capacity.
* Hip joint dysplasia.
* Sequelae to previous hip joint disorder in childhood.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04

PRIMARY OUTCOMES:
Acetabular component migration evaluated by RSA

SECONDARY OUTCOMES:
BMD in the surrounding bone of the acetabular implant

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD., Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital,, Aarhus, Denmark